CLINICAL TRIAL: NCT00026884
Title: Collection of Serum and Tissue Samples From Patients With Biopsy-Proved or Suspected Malignant Diseases
Brief Title: Collection of Serum and Tissue Samples From Patients With Biopsy-Proved or Suspected Malignant Disease
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970147; 97-C-0147; NCT00897585 (obsolete NCT alias)
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Malignant Neoplasms; Hereditary Neoplastic Syndromes; Kidney Cancer; Renal Cancer; Bladder Cancer
Keywords: Serum; Collection of Tissue; Malignant Disease; Molecular Basis; Genome Sequencing; Natural History
MeSH Terms: conditions — Neoplasms; Neoplastic Syndromes, Hereditary; Kidney Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family Members: Family members (related by blood) of patients who have or are suspected of having a malignant disease or an inherited genitourinary malignant disorder
- Patients: Patients with biopsy-proven malignant diseases; or patients suspected of having a malignant disease; or patients who have or who are suspected of having an inherited genitourinary malignant disorder

SUMMARY:
Selected patients suspected of having or with prior biopsy proof of malignant disease will be seen in the Urologic Oncology Branch, NCI. Blood samples may be collected at the time of the initial visit and at periodic intervals during the course of the disease. These samples will be stored in the tissue bank of the Urologic Oncology Branch. Aliquots of malignant and normal tissue will be collected at the time of surgery and stored in the tissue bank, Urologic Oncology Branch, NCI. These materials will be used in the research efforts of the Urologic Oncology Branch, NCI....

DETAILED DESCRIPTION:
Background

Kidney, prostate, bladder, testis and penile cancer account for 22% of cancers diagnosed in the United States and are responsible for 10% of cancer deaths each year in the U.S. Understanding the genes and gene pathways that cause genitourinary malignancies will provide the foundation for the development of targeted therapeutic agents for patients affected with these cancers. Since 1982 investigators in the Urologic Oncology Branch have been studying the genetic basis of urologic cancers. The identification of the genes for cancer of the kidney has led to the approval by the FDA of a number of new agents for patients with advanced disease. It is our goal to study the cancer gene pathways of genitourinary malignancies in order to further understand the cancer gene pathways that cause these diseases.

Objectives

Collection of benign and malignant tissue from patients with known or suspected cancer

Collection of benign and malignant tissue from patients with rare inherited conditions associated with an increased risk for kidney cancer

Determine the molecular genetic differences between normal and tumorigenic tissues

Investigate the categories of genes/ biochemical pathways such as those that influence the cell cycle, angiogenesis, metabolic changes, and metastatic potential

Examine protein expression and bioimmunoassays investigating potential genetic markers

Investigate cellular/biochemical response to existing and novel therapeutic agents.

Investigate quality of life in men who have prostate cancer

Investigate molecular genetic basis of urologic malignancies

Examine cell free DNA and circulating tumor DNA for cancer gene mutations

Eligibility

Patients with biopsy-proven malignant disease

Patients suspected of having malignant disease

Patients with known or suspected inherited urologic malignant disorder

Family members (related by blood) of patients who have or are suspected of having an inherited genitourinary disorder or malignancy

Family members of patients with a DNA variant

Design

Patients will be screened for eligibility in the Urologic Oncology Branch Clinic

Blood and urine samples may be obtained

Normal and malignant tissue may be collected from patients undergoing clinically indicated surgical procedures

Basic scientific research will be performed on collected specimens

Patients will have the option to be contacted if a result is detected that would affect their health and they will be given the opportunity to be evaluated and re-tested on an IRB approved protocol if available

Germline and somatic whole genome exome sequencing may be performed

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult and minor patients with biopsy-proven malignant disease
* Adult and minor patients suspected of having a malignant disease
* Patients who have or are suspected of having an inherited genitourinary malignant disorder
* Participants must be >= 2 years of age
* Family members (related by blood) of patients who have or are suspected of having a malignant disease or an inherited genitourinary malignant disorder.
* All patients and guardians, for children younger than 18 years of age, must sign an informed consent document indicating their understanding of the investigational nature and the risks of this study before any protocol related studies are performed. Patients under the age of 18 but who are age 13 or older will be asked to sign an assent document prior to participation.

EXCLUSION CRITERIA:

- Subjects whose co-morbidities preclude surgical intervention.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients with biopsy-proven malignant disease 2. Patients suspected of having malignant disease 3. Patients with known or suspected urologic malignant disorders who have clinically indicated urologic or non-urologic surgical lesion 4. Family members of patients suspected of having an inherited genitourinary malignancy 5. Family members of patients with a DNA variant
Sampling Method: Non-Probability Sample
Enrollment: 5950 (Estimated)
Dates: Start 1998-03-12 (Actual)

PRIMARY OUTCOMES:
Investigate quality of life in men who have prostate cancer. | on-going
  Prostate cancer patients that have improvement in quality of life
Investigate molecular genetic basis of urologic malignancies | on-going
  Investigate molecular genetic basis of urologic malignancies
Investigate cellular/biochemical response to existing and novel therapeutic agents. | on-going
  Collection of blood, urine, saliva, and/or benign and malignant tissue
Examine protein expression and bioimmunoassays investigating potential genetic markers. | on-going
  Detection and expression analysis of gene(s)
Determine the molecular genetic differences between normal and tumorigenic tissues. | on-going
  Molecular genetic differences between normal and tumorigenic tissues
Collection of benign and malignant tissue from patients with rare inherited conditions associated with an increased risk for kidney cancer. | on-going
  Collection of blood, urine, saliva, and/or benign and malignant tissue
Collection of benign and malignant tissue from patients with known or suspected cancer. | on-going
  Collection of blood, urine, saliva, and/or benign and malignant tissue

CONTACTS AND LOCATIONS:
Overall Officials: W. Marston Linehan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Merriman KM, Harmon SA, Belue MJ, Yilmaz EC, Blake Z, Lay NS, Phelps TE, Merino MJ, Parnes HL, Law YM, Gurram S, Wood BJ, Choyke PL, Pinto PA, Turkbey B. Comparison of MRI-Based Staging and Pathologic Staging for Predicting Biochemical Recurrence of Prostate Cancer After Radical Prostatectomy. AJR Am J Roentgenol. 2023 Dec;221(6):773-787. doi: 10.2214/AJR.23.29609. Epub 2023 Jul 5. PMID 37404084
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1997-C-0147.html